CLINICAL TRIAL: NCT06619912
Title: Dexmedetomidine in Reducing Postoperative Delirium in Cardiac Surgery Patients：a Single-center, Double- Blind, Controlled Trial
Brief Title: Dexmedetomidine in Reducing Postoperative Delirium in Cardiac Surgery Patients
Acronym: DREAMS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20242259
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Delirium; Preoperative Sleep Disorder
Keywords: postoperative delirium; preoperative sleep disorder; dexmedetomidine; cardiopulmonary coupling
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): The Dexmedetomidine group will receive dexmedetomidine nasal spray （1.5ug/kg, ideal body weight) at the night before surgery and 30 minutes before induction.
  Interventions: Drug: Dexmedetomidine nasal spray
- Control group (No Intervention): In the control group, the treatment is sodium chloride 0.9% nasal spray. Follows the same rules as in the experimental group.

INTERVENTIONS:
Drug: Dexmedetomidine nasal spray — Participants will be randomised to receive either dexmedetomidine or saline nasal spray (1.5ug/kg, ideal body weight) at the night before surgery and 30 minutes before induction.
  Arms: Dexmedetomidine group

SUMMARY:
Delirium is a common consequence of cardiac surgery and associates with poor outcomes. Multiple causes can trigger delirium occurence, and it has been hypothesised that sleep disturbances can be one of them. Dexmedetomidine may be effective in reducing delirium. The aim of this study was to demonstrate preoperative dexmedetomidine nasal spray in cardiac surgery patients can reduce postoperative delirium by improving preoperative sleep.

DETAILED DESCRIPTION:
Due to special reasons such as surgical trauma, irritability, extracorporeal circulation, the incidence of postoperative delirium (POD) after cardiovascular surgery ranges from 26% to 52%. POD is an acute organic brain syndrome characterised by cognitive impairment and alteration of consciousness. The implications of this acute form of brain injury are profound. Patients who experience delirium are more likely to experience increased short- and long-term mortality, decrease in long-term cognitive function, increase in hospital length of stay and increased complications of hospital care. Given the numerous adverse effects of POD, it is crucial to explore the mechanisms for the prevention and management of POD.

Dexmedetomidine (Dex) is a highly selective α 2-adrenergic receptor agonist that produces sedative and hypnotic effects by activating the α 2-adrenergic receptor in the brainstem locus coeruleus, and has a certain neuroprotective effect. In recent years, the prevention of postoperative delirium by Dex has been a hot topic in the field of anesthesia. However, recent studies have found contradictory conclusions on aforementioned topic.

The heterogeneity of the subject population may be the reason for the current contradictory conclusions. Tang et al. conducted a meta-analysis of all RCTs regarding perioperative sleep interventions and postoperative delirium, and found that in the subgroup where interventions effectively improved patients' sleep quality, the effect of reducing the incidence of postoperative delirium was more significant. At the same time, the incidence of delirium did not decrease in the subgroup where sleep quality was not improved. Sleep disorders play a crucial role in the pathogenesis of POD.

In this DREAMS study, we plan to conduct a single center double-blind randomized controlled trial involving patients undergoing extracorporeal circulation cardiac surgery to explore whether administering Dex nasal spray the night before surgery and 30 minutes before anesthesia induction can improve preoperative sleep quality and reduce the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Cardiac surgery with cardiopulmonary bypass.
3. Ability to provide consent.

Exclusion Criteria:

1. Preoperative schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, history of neurosurgery, or Mini-mental State Examination(MMSE) score: illiteracy<17, primary school level<20, high school level <24.
2. Patients with sick sinus syndrome, severe sinus bradycardia (heart rate<50 beats/minute), grade II or above atrioventricular block, and no pacemaker implanted.
3. Unable to communicate due to coma, severe dementia, or language barriers prior to surgery.
4. Patients with severe liver dysfunction (Child Pugh C grade), renal dysfunction (preoperative dialysis), ASA grade V or expected survival ≤ 24 hours.
5. Heart transplant surgery
6. Surgery for congenital heart disease.
7. Deep hypothermic circulatory arrest surgery.
8. Already enrolled in other study patients.
9. Refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium occurrence | within 1 week after operation
  Delirium occurrence was evaluated with confusion assessment method for the ICU(CAM- ICU) or 3-Minute Confusion Assessment Method (3D-CAM) two times per day during the 7 days following surgery.

SECONDARY OUTCOMES:
Delirium severity measurement | 1week after surgery
  Delirium severity is assessed using Confusion Assessment Method for the intensive care unit (CAM-ICU)-7, score 3-5 is considered as mild to moderate delirium, score 6-7 is considered as severe delirium
Delirium subtypes | 1week after surgery
  Hyperactive POD was defined as a RASS score of +1 to +4 accompanying a positive CAM-ICU/3D-CAM, hypoactive POD was defined as a RASS score of -3 to 0 accompanying a positive CAM-ICU/3D-CAM, mixed POD was defined by simultaneous or sequential exhibition of hypoactive and hyperactive manifestationscare unit (CAM-ICU)-7, score 3-5 is considered as mild to moderate delirium, score 6-7 is considered as severe delirium
Duration of delirium | 1week after surgery
  Duration of delirium is assessed using Confusion Assessment Method for the intensive care unit (CAM-ICU) or 3-Minute Confusion Assessment Method (3D-CAM)
Hospital length of stay. | From the date of surgery until the date patient discharge from hospital, assessed up to 30 days]
  Hospital length of stay.
In- hospital mortality | From the date of surgery until the date patient discharge from hospital, assessed up to 30 days]
  In- hospital mortality
NRS score of sleep during the first night after surgery | The first night after surgery
  NRS score of sleep during the first night after surgery
Postoperative anxiety and depression | 1week after surgery
  Postoperative anxiety and depression are assessed using Hospital Anxiety and Depression Scale (HADS)
Pain intensity | 1week after surgery
  1) Pain intensity is assessed using the NRS at rest and during movement daily for 7 postoperative days

OTHER OUTCOMES:
Postoperative occurence of AKI | 1week after surgery
  AKI occurrence was evaluated with KIDGO guideline during the 7 days following surgery.
Plasma concentration of pTau-217 | 24h after surgery
  Preoperative plasma pTau-217 level is detected after the second dose of the test drug is conducted, and the postoperative plasma pTau-217 level is detected 24 hours after surgery. Plasma pTau-217 level is determined using the Quanterix method that is based on ultrasensitive Simoa technology,on an HD-X analytical platform.
Postoperative occurence of atrial fibrillation | 1week after surgery
  Postoperative occurence of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, M.D., phd, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 12 months

REFERENCES:
- [Background] Wu M, Liang Y, Dai Z, Wang S. Perioperative dexmedetomidine reduces delirium after cardiac surgery: A meta-analysis of randomized controlled trials. J Clin Anesth. 2018 Nov;50:33-42. doi: 10.1016/j.jclinane.2018.06.045. Epub 2018 Jun 27. PMID 29958125
- [Background] Turan A, Duncan A, Leung S, Karimi N, Fang J, Mao G, Hargrave J, Gillinov M, Trombetta C, Ayad S, Hassan M, Feider A, Howard-Quijano K, Ruetzler K, Sessler DI; DECADE Study Group. Dexmedetomidine for reduction of atrial fibrillation and delirium after cardiac surgery (DECADE): a randomised placebo-controlled trial. Lancet. 2020 Jul 18;396(10245):177-185. doi: 10.1016/S0140-6736(20)30631-0. PMID 32682483